CLINICAL TRIAL: NCT03032250
Title: Prepare to Care, A Supported Self-Management Intervention for Head and Neck Cancer Caregivers
Brief Title: Prepare to Care, A Supported Self-Management Intervention for Head and Neck Cancer CaregiversHead and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00038084; NCI-2016-02045 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 99616 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH); R03CA208560 (NIH)
Record Dates: First submitted 2017-01-17; First posted 2017-01-26 (Estimated); Results first posted 2021-07-01 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Caregiver; Malignant Head and Neck Neoplasm; Paranasal Sinus Squamous Cell Carcinoma; Salivary Gland Squamous Cell Carcinoma; Stage I Hypopharyngeal Squamous Cell Carcinoma; Stage I Laryngeal Squamous Cell Carcinoma; Stage I Lip and Oral Cavity Squamous Cell Carcinoma; Stage I Oropharyngeal Squamous Cell Carcinoma; Stage II Hypopharyngeal Squamous Cell Carcinoma; Stage II Laryngeal Squamous Cell Carcinoma; Stage II Lip and Oral Cavity Squamous Cell Carcinoma; Stage II Oropharyngeal Squamous Cell Carcinoma; Stage III Hypopharyngeal Squamous Cell Carcinoma; Stage III Laryngeal Squamous Cell Carcinoma; Stage III Lip and Oral Cavity Squamous Cell Carcinoma; Stage III Oropharyngeal Squamous Cell Carcinoma; Stage IV Hypopharyngeal Squamous Cell Carcinoma; Stage IV Laryngeal Squamous Cell Carcinoma; Stage IV Lip and Oral Cavity Squamous Cell Carcinoma; Stage IV Oropharyngeal Squamous Cell Carcinoma; Stage IVA Hypopharyngeal Squamous Cell Carcinoma; Stage IVA Laryngeal Squamous Cell Carcinoma; Stage IVA Lip and Oral Cavity Squamous Cell Carcinoma; Stage IVA Oropharyngeal Squamous Cell Carcinoma; Stage IVB Hypopharyngeal Squamous Cell Carcinoma; Stage IVB Laryngeal Squamous Cell Carcinoma; Stage IVB Lip and Oral Cavity Squamous Cell Carcinoma; Stage IVB Oropharyngeal Squamous Cell Carcinoma; Stage IVC Hypopharyngeal Squamous Cell Carcinoma; Stage IVC Laryngeal Squamous Cell Carcinoma; Stage IVC Lip and Oral Cavity Squamous Cell Carcinoma; Stage IVC Oropharyngeal Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Lip and Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal SCC; Recurrent Paranasal Sinus Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Lymphoid Interstitial Pneumonia | interventions — Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I Supportive Care (Prepare to Care kit) (Experimental): Caregivers watch introduction video on a DVD over 10 minutes at baseline. Caregivers receive Prepare to Care kit including 8 workbook modules and complete at least 1 module over 30-45 minutes each week. Caregivers also attend interventionist session over 10-30 minutes weekly.
  Interventions: Other: Communication Intervention; Other: Watch video; Other: Module completion of the Prepare to Care kit; Other: Quality-of-Life Assessment; Other: Survey Administration; Other: Salivary cortisol collection
- Group II Control Group (Experimental): Caregivers received standard of care throughout course of intervention, with option to receive study intervention at end of study
  Interventions: Other: Watch video; Other: Module completion of the Prepare to Care kit; Other: Quality-of-Life Assessment; Other: Survey Administration; Other: Salivary cortisol collection

INTERVENTIONS:
Other: Communication Intervention — Attend interventionist sessions
  Arms: Group I Supportive Care (Prepare to Care kit)
Other: Watch video — Watch video on a DVD
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Module completion of the Prepare to Care kit — Complete modules of the Prepare to Care kit
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Ancillary studies
Other: Salivary cortisol collection — Obtained at three times a day (at awakening, 30 minutes post awakening and bedtime) for two consecutive days for eligible caregivers in both groups. Samples collected by placing a cotton ball under the tongue for approximately 1-2 minutes which is subsequently stored in a plastic tube and refrigerated.

SUMMARY:
This pilot clinical trial studies how well Prepare to Care kit works in improving caregiver support in patients with stage I-IV head and neck cancer that is new or has come back. Prepare to Care kit may increase knowledge about head and neck cancer and enhance stress-management skills.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess feasibility (accrual, participation, and retention) and acceptability of a supported self-management intervention for psycho-education and stress management skills building designed for informal caregivers (intervention group n=20; waitlist control group, n=20) of head and neck cancer (HNC) patients undergoing radiotherapy (RT).

II. To obtain preliminary data on caregiver intermediate (self-efficacy for [a] coping with cancer and [b] abbreviated progressive muscle relaxation) and outcome variables (burden, psychological distress, quality of life) in intervention caregivers and waitlist control caregivers at the start of radiation (T1), end of radiation (T2), and 6-weeks post-radiation (T3).

III. To compare intermediate (self-efficacy for (a) coping with cancer and (b) abbreviated progressive muscle relaxation) and outcome variables (burden, psychological distress, quality of life) between intervention caregivers and waitlist control caregivers at T1, T2, and T3.

IV. To obtain preliminary data on caregiver cortisol response (cortisol slope, cortisol awakening

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Caregivers watch introduction video on a digital video disc (DVD) over 10 minutes at baseline. Caregivers receive Prepare to Care kit including 8 workbook modules and complete at least 1 module over 30-45 minutes each week. Caregivers also attend interventionist session over 10-30 minutes weekly.

GROUP II: Caregivers receive educational intervention as in Group I but do not attend interventionist sessions.

ELIGIBILITY:
Inclusion Criteria:

CAREGIVERS:

* Providing the majority of the informal (unpaid) care during radiation therapy for a patient meeting inclusion criteria and participating in study

CARE-RECIPIENTS:

* Has a new or recurrent American Joint Committee on Cancer (AJCC) stage I-IV squamous cell carcinoma of the upper aerodigestive tract (including lip/oral cavity, nasopharynx, salivary gland, oropharynx, hypopharynx, paranasal sinus, and larynx cancers)
* Has planned external beam radiotherapy (+/- chemotherapy) for 6-7 weeks
* Has an informal (unpaid) caregiver during radiation therapy who is participating in study

Exclusion Criteria:

* CAREGIVERS: Has a current cancer diagnosis
* CAREGIVERS: Cannot read/communicate in English
* CAREGIVERS: Have an endocrine disorder (e.g., diabetes and thyroid disorders), or is currently taking a steroid based medication will not be eligible to participate in the saliva portion of the study
* CARE-RECIPIENTS: Cannot read/communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandylen Nightingale, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Nightingale C, Sterba KR, Levine B, Tooze JA, Greven K, Frizzell B, Hughes RT, Snavely A, Lesser GJ, Norona S, Pleasant K, Weaver KE. Feasibility and Acceptability of a Multi-Modality Self-Management Intervention for Head and Neck Cancer Caregivers: A Pilot Randomized Trial. Integr Cancer Ther. 2022 Jan-Dec;21:15347354221098984. doi: 10.1177/15347354221098984. PMID 35575280

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I Supportive Care (Prepare to Care Kit) | Group II Control Group
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group II Control Group: Caregivers received standard of care throughout course of intervention, with option to receive study intervention at end of study."
  Watch video: Watch video on a DVD
  Module completion of the Prepare to Care kit: Complete modules of the Prepare to Care kit
  Quality-of-Life Assessment: Ancillary studies
  Survey Administration: Ancillary studies
  Salivary cortisol collection: Obtained at three times a day (at awakening, 30 minutes post awakening and bedtime) for two consecutive days for eligible caregivers in both groups. Samples collected by placing a cotton ball under the tongue for approximately 1-2 minutes which is subsequently stored in a plastic tube and refrigerated.
- Total: Total of all reporting groups
Arm/Group | Group I Supportive Care (Prepare to Care Kit) | Group II Control Group | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (15.5) | 57.4 (11.8) | 56.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 4 | 21
  Male | 0 | 14 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 18 | 34
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 16 | 13 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Noting Quite a Bit/Very Much Helpful to Survey Questions
Description: 10-item quantitative survey will be developed for study to assess how much caregivers liked different aspects of the intervention. Acceptability will be summarized quantitatively and qualitatively. These acceptability questions were asked only of caregivers in the intervention group - Group 1 Supportive Care (Prepare to Care Kit). All data is based on participants answering the acceptability questions as "Quite a Bit/Very Much Helpful" for the intervention materials. Not all participants answered this part of the outcome measure.
Time Frame: Six weeks post radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Group I Supportive Care (Prepare to Care Kit)
Number analyzed (Participants) | 17
Participants
  Introductory DVD | 4
  Meetings with study interventionist | 6
  Relaxation CD | 7
  Weekly text reminders | 6
  Weekly email reminders | 4
  Study website | 0
  Clinic iPads | 0
  Cancer Education workbook | 9
  Utilizing Resources workbook | 7
  Managing Time workbook | 7
  Seeking/Accepting Support workbook | 7
  Communicating with Others workbook | 7
  Healthy Behaviors workbook | 7
  Positive Coping workbook | 7
  Muscle Relaxation workbook | 7

2. Primary Outcome: Accrual Assessed by Number of Caregivers Who Agreed to Participate Divided by the Number of Months of Recruitment
Description: 38 patient/caregiver dyads agreed to participate, 22 months of recruitment, for accrual rate of 1.7 (caregiver) participants per month
Time Frame: Up to 1 year
Population: 38 patient/caregiver dyads agreed to participate, 22 months of recruitment, for accrual rate of 1.7 (caregiver) participants per month
Measure: Number; unit: participants/months
Groups:
- All Participants: Caregivers watch introduction video on a DVD over 10 minutes at baseline. Caregivers receive Prepare to Care kit including 8 workbook modules and complete at least 1 module over 30-45 minutes each week. Caregivers also attend interventionist session over 10-30 minutes weekly.
  Communication Intervention: Attend interventionist sessions
  Watch video: Watch video on a DVD
  Module completion of the Prepare to Care kit: Complete modules of the Prepare to Care kit
  Quality-of-Life Assessment: Ancillary studies
  Survey Administration: Ancillary studies
  Salivary cortisol collection: Obtained at three times a day (at awakening, 30 minutes post awakening and bedtime) for two consecutive days for eligible caregivers in both groups. Samples collected by placing a cotton ball under the tongue for approximately 1-2 minutes which is subsequently stored in a plastic tube and refrigerated.
Arm/Group | All Participants
Number analyzed (Participants) | 38
participants/months | 1.7

3. Primary Outcome: Change in Caregiver Burden Assessed by Caregiver Reaction Assessment (CRA)
Description: 21-item instrument assessing positive and negative aspects of caregiving (esteem, lack of family support, finances, schedule, and health). The CRA has been tested in cancer caregivers; demonstrated validity and reliability. Minimum and maximum scoring scale: BASELINE: Scores for esteem 15-31; lack of family support 5-15, impact of finances 3-12, impact of schedule 12-23, impact of health 11-16). AFTER RADIOTHERAPY: Scores for esteem 20-31; lack of family support 9-17, impact of finances 7-11, impact of schedule 14-22, impact of health 12-17). The higher the score the more the item being assessed impacted the participant.
Time Frame: Baseline and following radiotherapy, assessed up to 1 year
Population: Not all participants submitted information after completion of radiotherapy.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group II No Interventionist Sessions: Caregivers receive educational intervention as in Group I but do not attend interventionist sessions
  Watch video: Watch video on a DVD
  Module completion of the Prepare to Care kit: Complete modules of the Prepare to Care kit
  Quality-of-Life Assessment: Ancillary studies
  Survey Administration: Ancillary studies
  Salivary cortisol collection: Obtained at three times a day (at awakening, 30 minutes post awakening and bedtime) for two consecutive days for eligible caregivers in both groups. Samples collected by placing a cotton ball under the tongue for approximately 1-2 minutes which is subsequently stored in a plastic tube and refrigerated.
Arm/Group | Group I Supportive Care (Prepare to Care Kit) | Group II No Interventionist Sessions
Number analyzed (Participants) | 17 | 18
score on a scale
  Esteem at baseline | 25.98 (3.6) | 25.88 (3.8)
  Lack of family support at baseline | 11.29 (2.69) | 11.25 (2.67)
  Impact on finances at baseline | 8.29 (2.28) | 8.89 (1.78)
  Impact on schedule at baseline | 17.35 (3.31) | 16.78 (4.1)
  Impact on health at baseline | 13.94 (1.48) | 13.67 (1.65)
  Esteem after radiotherapy: number analyzed (Participants) | 12 | 16
  Esteem after radiotherapy | 25.75 (3.31) | 25.30 (4.19)
  Lack of family support after radiotherapy: number analyzed (Participants) | 12 | 16
  Lack of family support after radiotherapy | 12.58 (2.23) | 11.19 (3.23)
  Impact on finances after radiotherapy: number analyzed (Participants) | 12 | 16
  Impact on finances after radiotherapy | 8.42 (1.16) | 8.25 (1.24)
  Impact on schedule after radiotherapy | 18.33 (2.74) | 16.56 (4.43)
  Impact on health after radiotherapy | 14.33 (1.61) | 14.38 (1.59)

4. Primary Outcome: Change in Psychological Distress - Center for Epidemiological Studies Depression (CESD)
Description: The score is the sum of the 20 questions. Possible scoring range is 0-60. A score of 16 points or more is considered depressed.
Time Frame: Before and after radiotherapy, assessed up to 1 year
Population: Not all participants completed this intervention after radiotherapy timeframe indicated for this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I Supportive Care (Prepare to Care Kit) | Group II No Interventionist Sessions
Number analyzed (Participants) | 17 | 18
score on a scale
  Score at baseline | 19.71 (13.05) | 19.28 (12.97)
  Score after radiotherapy: number analyzed (Participants) | 12 | 16
  Score after radiotherapy | 19.00 (15.66) | 13.58 (8.65)

5. Primary Outcome: Change in Quality of Life Assessed by Caregiver Quality of Life Index-Cancer (CqoL-Canc)
Description: 35-item instrument assessing dimensions of caregiver quality of life (burden, disruptiveness, positive adaptation, financial concerns). The Cqol-Canc has demonstrated validity and reliability. Minimum and maximum score at baseline is a range of 9-78 and after radiotherapy a range of 2-73. The higher the score the greater the level of change in the quality of life for participants.
Time Frame: Before and after radiotherapy, assessed up to 1 year
Population: Not all participants completed this intervention after radiotherapy as indicated for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I Supportive Care (Prepare to Care Kit) | Group II No Interventionist Sessions
Number analyzed (Participants) | 17 | 17
score on a scale
  At baseline | 87.63 (25.95) | 87.26 (20.32)
  After radiotherapy: number analyzed (Participants) | 12 | 16
  After radiotherapy | 92.55 (22.09) | 89.86 (18.78)

6. Primary Outcome: Frequency of Intervention Modules Utilized Assessed by Caregiver Logs
Description: Data on intervention resources used and time spent using them based on caregivers in intervention group
Time Frame: Up to 1 year
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group I Supportive Care (Prepare to Care Kit)
Number analyzed (Participants) | 17
Minutes
  Cancer Education | 22.3 (10.2)
  Utilizing Resources | 38.7 (20.1)
  Seeking/ Accepting Support | 55.2 (27.8)
  Communicating with others | 40.3 (12.7)
  Managing Time | 40.8 (26.9)
  Coping | 66.7 (51.1)
  Practicing Healthy Behaviors | 48 (15.6)
  Relaxation CD | 58 (18.1)

7. Primary Outcome: Number of Participants in Agreement to Perform Interventions
Description: Participation assessed by number of eligible participants who agreed to participate and complete study interventions.
Time Frame: Up to 1 year
Population: 90 eligible patient/caregiver dyads, 38 agreed to participate
Measure: Count of Participants; unit: Participants
Groups:
- Combination of Intervention and Control Groups to Assess Participation: Participation assessed by proportion of eligible participants who agreed to participate
Arm/Group | Combination of Intervention and Control Groups to Assess Participation
Number analyzed (Participants) | 90
Participants | 38

8. Primary Outcome: Retention Assessed by Number of Participants Who Completed the End of Radiotherapy Visit Divided by the Number Who Agreed to Participate
Time Frame: Up to 1 year
Population: 38 agreed to participate (19 in caregiver intervention group, 19 in caregiver control group)
Measure: Count of Participants; unit: Participants
Arm/Group | Group I Supportive Care (Prepare to Care Kit) | Group II No Interventionist Sessions
Number analyzed (Participants) | 38 | 38
Participants | 12 | 16

9. Primary Outcome: Self-efficacy in Abbreviated Progressive Muscle Relaxation (APMR)
Description: A 3-item instrument developed for study to evaluate self-efficacy in APMR. Minimum to maximum scores range from 3-27. Higher scores demonstrate higher self efficacy in participants.
Time Frame: At baseline and up to the end of radiotherapy, assessed up to 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I Supportive Care (Prepare to Care Kit) | Group II No Interventionist Sessions
Number analyzed (Participants) | 17 | 18
score on a scale
  At baseline | 11.88 (6.53) | 13.33 (5.36)
  After radiotherapy | 16.08 (2.68) | 12.19 (5.59)

10. Primary Outcome: Self-efficacy in Coping With Cancer Caregiver Inventory
Description: 21-item instrument assessing caregivers' perceived self-efficacy for coping with cancer (managing medical information, caring for care recipient, caring for oneself, managing difficult interactions/emotions); demonstrated validity and reliability. Minimum and maximum scores range from 10-63. Higher scores indicate higher self-efficacy in coping with cancer from the participants.
Time Frame: At baseline and up to the end of radiotherapy, assessed up to 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I Supportive Care (Prepare to Care Kit) | Group II No Interventionist Sessions
Number analyzed (Participants) | 17 | 18
score on a scale
  Managing medical information at baseline | 22.35 (3.26) | 22.00 (3.29)
  Caring for care recipient at baseline | 52.94 (9.65) | 55.11 (6.11)
  Caring for oneself at baseline | 25.71 (10.44) | 28.06 (7.83)
  Managing difficult interactions/emotions at baseline | 34.52 (10.96) | 39.13 (7.95)
  Managing medical information after radiotherapy | 23.08 (2.54) | 22.43 (4.80)
  Caring for care recipient after radiotherapy | 54.42 (5.62) | 54.98 (6.82)
  Caring for oneself after radiotherapy | 25.75 (9.40) | 31.30 (8.26)
  Managing difficult interactions/emotions after radiotherapy | 37.92 (10.03) | 39.68 (7.86)

11. Other Pre Specified Outcome: Salivary Cortisol Collection
Description: For eligible caregivers only - collected three times a day (at awakening, 30 minutes post-awakening, and bedtime) for two consecutive days following T1 (start of radiation), T2 (end of radiation), and T3 (6 weeks post radiation). To obtain preliminary data on caregiver cortisol response (cortisol slope, cortisol awakening response, area under the curve, and intra-individual cortisol variability). Investigators will use a mixed model to evaluate differences between the groups in these parameters at times T1 and T2 and T3
Time Frame: Up to 1 year
Population: Analysis of this outcome measure is currently incomplete and cannot be reported as this time as the information is not available.
Arm/Group | Group I Supportive Care (Prepare to Care Kit) | Group II Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Group I Supportive Care (Prepare to Care Kit) | Group II Control Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT03032250/Prot_SAP_000.pdf
  • Informed Consent Form: Caregiver Informed Consent (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT03032250/ICF_001.pdf
  • Informed Consent Form: Patient Informed Consent (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT03032250/ICF_002.pdf